CLINICAL TRIAL: NCT01768936
Title: Procalcitonin Ratio's Impact on the Decision Upon On-demand Relaparotomy in Septic Peritonitis
Status: Completed | Type: Observational
Sponsor: CHIR-Net (Network)
Responsible Party: Sponsor
Other Study IDs: TUM-PCT-1; PCTRatio Reevaluation (Other: CHIR-Net)
Record Dates: First submitted 2013-01-10; First posted 2013-01-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Secondary Peritonitis After Intestinal Perforation
Keywords: on-demand relaparotomy; PCT; procalcitonin; peritonitis; sepsis; focus index
MeSH Terms: conditions — Peritonitis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- eliminated infectious abdominal focus
- persisting/progressing infectious abdominal focus

SUMMARY:
Procalcitonin (PCT) serum levels are monitored in patients with secondary peritonitis after initial operative focus elimination to investigate the PCT ratio's impact on decision-making for or against early relaparotomy in the on-demand relaparotomy concept of secondary septic peritonitis.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* necessity for operative intervention to eliminate an infectious peritoneal / abdominal focus after organ perforation
* abdominal sepsis according to the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference definition

Exclusion Criteria:

* pregnancy
* immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive postoperative surgical patients on ICU after intestinal perforation or anastomotic leakage with indication for surgical focus elimination
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
prediction of focus elimination: cured patients versus patients with persisting peritonitis (definitions see below) | participants will be followed for the duration of hospital stay, an expected average of 21 days
  definition of 'focus elimination': patients with intestinal perforation or anastomotic leakage develop (local) peritonitis and consecutive abdominal sepsis. These patients need surgical intervention for focus elimination. This operative intervention aims to eradicate all infectious material and is intended to remove the leaking intestinal lesion. Whether this focus is eliminated or not can be controlled by either planned relaparotomy (normally within 48h after the first operation) or on demand relaparotomy in case of clinical deterioration. The focus can be assumed to be eliminated in all cases where either relaparotomy reveals no ongoing infection or persisting focus and whenever a patient recovers rapidly after initial surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar der TU München, Munich, Germany